CLINICAL TRIAL: NCT06725290
Title: Digital Assessment of Dry Eye Diseases in Acne Vulgaris Patients Receiving Isotretinoin Therapy
Brief Title: Dry Eye Disease With Isotretinoin ISOTRETINOIN
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hagar El Sayed, University doctor, Cairo University
Other Study IDs: Dry eye with isotretinoin
Record Dates: First submitted 2024-12-08; First posted 2024-12-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low dose isotretinoin: Acne patients taking 20 mg daily isotretinoin
  Interventions: Diagnostic Test: Ocular Surface Disease Index (OSDI) questionnaire
- high dose isotretinoin: Acne patients taking 0.5 mg/kg daily dose of isotretinoin
  Interventions: Diagnostic Test: Ocular Surface Disease Index (OSDI) questionnaire
- Normal control
  Interventions: Diagnostic Test: Ocular Surface Disease Index (OSDI) questionnaire

INTERVENTIONS:
Diagnostic Test: Ocular Surface Disease Index (OSDI) questionnaire — The OSDI is a validated, self-administered questionnaire for assessing the presence and severity of ocular surface disease symptoms. The OSDI questionnaire includes 12 questions about the respondent's past week experience with the ocular symptoms, vision-related function, and environmental triggers

SUMMARY:
The study aims to explore the effects of isotretinoin therapy on the dry eye parameters in acne vulgaris patients & determine if it is dose-dependent or not.

DETAILED DESCRIPTION:
To measure the tear film, the eye lid thickness, the meibomian gland function and to do objective tests for comparison

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe acne on isotretinoin

Exclusion Criteria:

* Occular diseases causing dry eye
* Pregnant females

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acne patients on isotretinoin
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Total ocular surface disease index (OSDI) SCORE | 3 months
  Total OSDI score ranged from 0 to 100 with means greater symptom severity